CLINICAL TRIAL: NCT04508543
Title: Assessing Patient-provider Interactions During the Preoperative Anesthesia Consult
Acronym: IMPLICIT
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brandon M Togioka, Principal Investigator, Oregon Health and Science University
Other Study IDs: Study00022536
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Racism; Healthcare Disparities; Minority Health
Keywords: Implicit Bias; Unconscious Bias; Racial disparities; Non-verbal communication; Anesthesia
MeSH Terms: conditions — Racism; Bias, Implicit; Nonverbal Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minority (Case): Self-identified as being a member of group traditionally underrepresented in the medical profession relative to the proportion in the general population: African-American/Black, Mexican-American, Native American (American Indians, Alaska Natives, and Native Hawaiians), and mainland Puerto Rican.
  Interventions: Other: Non-verbal communication score
- Caucasian (Control): Self-identified as Caucasian and Non-Hispanic
  Interventions: Other: Non-verbal communication score

INTERVENTIONS:
Other: Non-verbal communication score — 1. To compare nonverbal communication score (NCS, range 0 - 4) between minority and Caucasian non-Hispanic patients. The score is a sum of four components, each contribute to a score range 0 - 1. The four components are: percent time spent with open body language, percent time spent interacting with the patient or surrogate, distance from the patient along the long axis of the patient's body (distance from the head), and distance from the patient along the axis perpendicular to the patient's body (distance from the handrail).

SUMMARY:
This will be a prospective, observational, single-center study to evaluate the effect of race and ethnicity on anesthesia provider-patient interactions. The investigators will also attempt to validate a new tool for assessing non-verbal communication during the preanesthesia consult.

Masking:

1. Patient
2. Anesthesia providers (attending anesthesiologist and resident or Certified Registered Nurse Anesthetist)

The patient and anesthesia provider(s) will not be told that the purpose of the study is to compare provider-patient interactions with minority patients to provider-patient interactions with Caucasian patients. The patient and anesthesia provider will be told that the investigators are conducting a study to evaluate provider-patient communication in the preanesthesia setting. The outcome assessor will be part of the research team. Accordingly, they will not be masked.

This is a pilot study void of sample size calculations. The investigators hope to enroll 100-200 patients in the study. While not a randomized study, the investigators hope to achieve a balanced number of minority and Caucasian patients.

DETAILED DESCRIPTION:
Primary Objective:

1. To compare nonverbal communication score (NCS, range 0 - 4) between minority and Caucasian non-Hispanic patients. The score is a sum of four components, each contribute to a score range 0 - 1. The four components are: percent time spent with open body language, percent time spent interacting with the patient or surrogate, distance from the patient along the long axis of the patient's body (distance from the head), and distance from the patient along the axis perpendicular to the patient's body (distance from the handrail).

Secondary Objectives:

1. To evaluate the association between NCS and patient medical risk, defined by the Charlson Co-Morbidity Index, range 0 - 37).
2. To evaluate the association between NCS and surgical risk. High risk surgeries will include intraperitoneal, intrathoracic, and suprainguinal vascular surgery, as classified by the Revised Cardiac Risk Index (RCRI). Lower risk surgery will include surgery in all other locations.
3. To evaluate the association between NCS and anesthesia decision making. In particular the investigators will evaluate the association between NCS and the incidence of arterial line insertion, the incidence of 2nd peripheral intravenous line insertion, the incidence of foley catheterization, the incidence of regional anesthesia blocks placed for postoperative analgesia, and parenteral morphine equivalent administration during surgery.
4. To evaluate the association between NCS and change in patient anxiety, as assessed by change in patient anxiety measured by the difference in anxiety on a Visual Analog Scale (VAS) score before preanesthesia anesthesia consult and after preanesthesia anesthesia consult.
5. To evaluate the association between NCS and the duration of the preanesthesia anesthesia consult, defined between the time the anesthesia provider enters the Post-Anesthesia Care Unit (PACU) bay and the time the anesthesia provider leaves the PACU bay.
6. To evaluate the impact of the observer to the study result, which will be assessed by recording the number of times the anesthesia provider looks at the outcome assessor.

Feasibility assessment: Feasibility for future investigation will be assessed by analyzing the following outcomes. Success will need to be found in all of the following areas to conclude a larger prospective study is feasible.

1. Is data collection by an observer technically feasible? Ability to obtain complete data to compute the primary outcome in > 95% of patients will be threshold for success.
2. Is the patient consent rate reasonable? Ability to consent > 50% of eligible patients will be the threshold for success.
3. Is there good agreement between raters? Mean NCS < 10% between raters will be the threshold for success.
4. Is the sample size, based upon the found difference in NCS between minority and Caucasian non-Hispanic patients, reasonable?

A sample size calculation yielding less than 500 patients will be the threshold for success.

Population: Patients will be 18 years old or greater, undergoing surgery in the South Operating Rooms at Oregon Health & Science University and possessing the capacity for consent.

Number of Sites: Single center trial

Study Arms: Minority (case): Self-identified as being a member of group traditionally underrepresented in the medical profession relative to the proportion in the general population: African-American/Black, Mexican-American, Native American (American Indians, Alaska Natives, and Native Hawaiians), and mainland Puerto Rican.

Control: Self-identified as Caucasian and non-Hispanic

Study Duration: Institutional Review Board submission and approval is expected to take 3 months. Study initiation, enrollment, and data collection is expected to take 12 months. Data analysis, manuscript writing, editing, submission and revision to a peer-reviewed journal is expected to take 12 months.

In summary, the study should be completed in under 3 years.

Subject Participation Duration: Individual subjects will be included the study for a portion of their time in the PACU for preanesthesia assessment. Total time of subject participation including time for recruitment, enrollment, data collection during the preanesthesia consult, and post-consult data collection will be less than 1 hour.

Estimated Time to Complete Enrollment: Estimated time from enrollment into study of the first subject to enrollment into study of the last subject is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Having surgery in the South Operating Rooms of Oregon Health & Science University
* Possessing the capacity for consent

Exclusion Criteria:

* Children
* Vulnerable populations including prisoners and decisionally impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients greater than or equal to 18 years old or greater, undergoing surgery and/or a surgical procedure in the South Operating Rooms at Oregon Health & Science University and possessing the capacity for consent, including minorities and Women of all racial/ethnic groups.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Nonverbal Communication Score (NCS score, range 0-4) | 1 hour
  The score is a sum of four components, each contribute to a score range 0 - 1.
  1) Percent time spent with open body language: defined as the anesthesia provider facing the patient and not placing anything between the anesthesia provider and the patient. 2) Percent time spent interacting with the patient or surrogate: Time spent interacting with the patient is defined as time the physician made eye contact with the patient or surrogate. Time spent talking to the patient, but not making eye contact will not be counted. Eye contact made during the physical examination will be counted. 3) Distance from the patient along the long axis of the patient's body (distance from the head) which will be assessed 15 seconds after the physician enters the preanesthesia bay. 4) Distance from the patient along the axis perpendicular to the patient's body (distance from the handrail).

SECONDARY OUTCOMES:
Non-Verbal Communication and Patient Medical Risk | 8 hours
  To evaluate the association between NCS and patient medical risk, defined by the Charlson Co-Morbidity Index, range 0 - 37).
NCS and Surgical Risk | 8 hours
  To evaluate the association between NCS and surgical risk. High risk surgeries will include intraperitoneal, intrathoracic, and suprainguinal vascular surgery, as classified by the Revised Cardiac Risk Index. Lower risk surgery will include surgery in all other locations.
Anesthesia Provider Observes Outcome Assessor | 8 hours
  To evaluate the impact of the observer to the study result, which will be assessed by recording the number of times the anesthesia provider looks at the outcome assessor.

OTHER OUTCOMES:
Evaluate following based on Non-Verbal Communication and Anesthesia Decision Making | 8 hours
  To evaluate the association between NCS and anesthesia decision making. In particular the investigators will evaluate the association between NCS and the incidence of the following procedures:
  1. Insertion of arterial line insertion,
  2. Insertion of second peripheral intravenous line
  3. Insertion of foley catheterization
  4. Nerve block placed for postoperative analgesia
Total Parenteral Morphine Equiv. Administered | 8 hours
  To evaluate the association between NCS and parenteral morphine equivalent administration during surgery.
Duration of Preanesthesia Anesthesia Consult | 1 hour
  To evaluate the association between NCS and the duration of the preanesthesia anesthesia consult, defined between the time the anesthesia provider enters the Post-Anesthesia Care Unit (PACU) bay and the time the anesthesia provider leaves the PACU bay.
Anxiety Measure | 8 hours
  To evaluate the association between NCS and change in patient anxiety, as assessed by change in patient anxiety measured by the difference in anxiety on a Visual Analog Scale (VAS) score before preanesthesia anesthesia consult and after preanesthesia anesthesia consult.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FitzGerald C, Hurst S. Implicit bias in healthcare professionals: a systematic review. BMC Med Ethics. 2017 Mar 1;18(1):19. doi: 10.1186/s12910-017-0179-8. PMID 28249596
- [Background] Elliott AM, Alexander SC, Mescher CA, Mohan D, Barnato AE. Differences in Physicians' Verbal and Nonverbal Communication With Black and White Patients at the End of Life. J Pain Symptom Manage. 2016 Jan;51(1):1-8. doi: 10.1016/j.jpainsymman.2015.07.008. Epub 2015 Aug 20. PMID 26297851
- [Background] Hall WJ, Chapman MV, Lee KM, Merino YM, Thomas TW, Payne BK, Eng E, Day SH, Coyne-Beasley T. Implicit Racial/Ethnic Bias Among Health Care Professionals and Its Influence on Health Care Outcomes: A Systematic Review. Am J Public Health. 2015 Dec;105(12):e60-76. doi: 10.2105/AJPH.2015.302903. Epub 2015 Oct 15. PMID 26469668
- [Background] Sabin J, Nosek BA, Greenwald A, Rivara FP. Physicians' implicit and explicit attitudes about race by MD race, ethnicity, and gender. J Health Care Poor Underserved. 2009 Aug;20(3):896-913. doi: 10.1353/hpu.0.0185. PMID 19648715
- [Background] AAMC. Percentage of all active physicians by race/ethnicity, 2018. Association of American Medical Colleges. https://www.aamc.org/data-reports/workforce/interactive-data/figure-18-percentage-all-active-physicians-race/ethnicity-2018. Published 2019. Accessed April 6, 2020, 2020.
- [Background] AAMC. Underrepresented in Medicine Definition. Association of American Medical Colleges. https://www.aamc.org/what-we-do/mission-areas/diversity-inclusion/underrepresented-in-medicine. Published 2004. Accessed March 10, 2020, 2020.
- [Background] Hagiwara N, Slatcher RB, Eggly S, Penner LA. Physician Racial Bias and Word Use during Racially Discordant Medical Interactions. Health Commun. 2017 Apr;32(4):401-408. doi: 10.1080/10410236.2016.1138389. Epub 2016 Jun 16. PMID 27309596
- [Background] Hagiwara N, Mezuk B, Elston Lafata J, Vrana SR, Fetters MD. Study protocol for investigating physician communication behaviours that link physician implicit racial bias and patient outcomes in Black patients with type 2 diabetes using an exploratory sequential mixed methods design. BMJ Open. 2018 Oct 18;8(10):e022623. doi: 10.1136/bmjopen-2018-022623. PMID 30341127
- [Background] Blair IV, Steiner JF, Fairclough DL, Hanratty R, Price DW, Hirsh HK, Wright LA, Bronsert M, Karimkhani E, Magid DJ, Havranek EP. Clinicians' implicit ethnic/racial bias and perceptions of care among Black and Latino patients. Ann Fam Med. 2013 Jan-Feb;11(1):43-52. doi: 10.1370/afm.1442. PMID 23319505
- [Background] Penner LA, Dovidio JF, Gonzalez R, Albrecht TL, Chapman R, Foster T, Harper FW, Hagiwara N, Hamel LM, Shields AF, Gadgeel S, Simon MS, Griggs JJ, Eggly S. The Effects of Oncologist Implicit Racial Bias in Racially Discordant Oncology Interactions. J Clin Oncol. 2016 Aug 20;34(24):2874-80. doi: 10.1200/JCO.2015.66.3658. Epub 2016 Jun 20. PMID 27325865
- [Background] Maina IW, Belton TD, Ginzberg S, Singh A, Johnson TJ. A decade of studying implicit racial/ethnic bias in healthcare providers using the implicit association test. Soc Sci Med. 2018 Feb;199:219-229. doi: 10.1016/j.socscimed.2017.05.009. Epub 2017 May 4. PMID 28532892
- [Background] Schulman KA, Berlin JA, Harless W, Kerner JF, Sistrunk S, Gersh BJ, Dube R, Taleghani CK, Burke JE, Williams S, Eisenberg JM, Escarce JJ. The effect of race and sex on physicians' recommendations for cardiac catheterization. N Engl J Med. 1999 Feb 25;340(8):618-26. doi: 10.1056/NEJM199902253400806. PMID 10029647
- [Background] Haider AH, Schneider EB, Sriram N, Dossick DS, Scott VK, Swoboda SM, Losonczy L, Haut ER, Efron DT, Pronovost PJ, Lipsett PA, Cornwell EE 3rd, MacKenzie EJ, Cooper LA, Freischlag JA. Unconscious race and social class bias among acute care surgical clinicians and clinical treatment decisions. JAMA Surg. 2015 May;150(5):457-64. doi: 10.1001/jamasurg.2014.4038. PMID 25786199
- [Background] Goyal MK, Johnson TJ, Chamberlain JM, Casper TC, Simmons T, Alessandrini EA, Bajaj L, Grundmeier RW, Gerber JS, Lorch SA, Alpern ER; Pediatric Care Applied Research Network (PECARN). Racial and Ethnic Differences in Antibiotic Use for Viral Illness in Emergency Departments. Pediatrics. 2017 Oct;140(4):e20170203. doi: 10.1542/peds.2017-0203. Epub 2017 Sep 5. PMID 28872046
- [Derived] Obeidat SS, Rakshe S, Fareh R, Norris K, Ye S, Zuo LW, Togioka BM. Impact of Unconscious Race Bias Among Anesthesia Providers on Nonverbal Communication During the Preoperative Anesthesia Consult: A Prospective, Observational Study. J Racial Ethn Health Disparities. 2025 Aug 22. doi: 10.1007/s40615-025-02604-5. Online ahead of print. PMID 40844570